CLINICAL TRIAL: NCT05269758
Title: Feasibility and Impact of an Activity-based Intervention for Strengthening Ingestive Functions in Elders With Sarcopenic Dysphagia: a Multiple-case Study
Brief Title: Feasibility and Impact of Resistance Training for Sarcopenic Dysphagia
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Tina Hansen, PhD, MSc.OT, Senior Researcher, Hvidovre University Hospital
Other Study IDs: H-19039031
Record Dates: First submitted 2022-02-04; First posted 2022-03-08 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Sarcopenia; Dysphagia
Keywords: Dysphagia; Sarcopenia; Resistance training; Task-oriented; Skill-based
MeSH Terms: conditions — Sarcopenia; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: activity-based resistance training of ingestive skills (ACT-ING-program) — The ACT-ING program is based on a task-oriented approach within motor behavior theories and combines resistance training principles with goal-directed and task-specific swallowing exercises in eating and drinking activities through a client-centered procedure informed by self-determination theory.

SUMMARY:
The purpose of the study is to test and optimize the feasibility of an activity-based resistance training program for patients with sarcopenic dysphagia. The study is a feasibility study designed as a multiple-case study with quantitative and qualitative data sources related to a number of feasibility outcomes and clinical outcomes during and after the intervention. Participants are 15 patients> 65 years of age are referred for dysphagia assessment by an Occupational Therapist (patients may be admitted to several different wards (endocrinology, pulmonary medicine, infectious medicine, gastrology). The intervention is offered during hospitalization and after discharge for a maximum of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Speaks and understand Danish language, and able to provide written informed consent for participation
* Dysphagia verified by a Gugging Swallowing Screen
* Generalized sarcopenia determined by a Danish version of the questionnaire SARC-F
* Sarcopenia of the swallowing mechanism indicated by reduced tongue strength measured with the Iowa Oral Performance Instrument

Exclusion Criteria:

* Dysphagia related to the esophagus
* Psychiatric diagnosis
* Neurodegenerative disease or
* Needs palliative care
* Admitted to hospital from a nursing home.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants admitted to an acute hospital for medical reasons (endocrinology, pulmonary medicine, infectious medicine, gastrology), and referred for dysphagia assessment by an Occupational Therapist .
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Intervention tolerance | During two therapy sessions per week in 12 weeks
  Time-series of participants rated level of concern for aspiration on a 100 mm VAS-scale ((left side = no concerns and right side = maximal concerns). The success criterion is that 80% of the VAS scales are in the area of 'no concerns' for aspiration.
Adverse effects | During two therapy sessions per week in 12 weeks
  Any expected and unintended events during the therapy sessions and the self-training are recorded.
Intervention usefulness | Up to 12 weeks
  Participant self-report on the subscale 'Value/usefulness' from the Intrinsic Motivation Inventory (IMI). The subscale covers 7 items to be rated on a 7-point Likert scale (1=Not at all true to 7=very true). A high score indicate high usability.
Acceptability | Up to 12 weeks
  Semi-structured interviews based on the Theoretical Framework of Acceptability

SECONDARY OUTCOMES:
Emotional wellbeing and global quality of life | Baseline and up to 12 weeks
  Two single VAS items using a horizontal line from 0 (worst imaginable emotional well-being / worst imaginable quality of life) to 100 mm (perfect emotional wellbeing /perfect quality of life).
Mealtime performance | Baseline and up to 12 weeks
  The McGill Ingestive Skills Assessment-version 2 (MISA2). The total score range from 36-108, where higher score indicate higher performance
Functional oral intake | Baseline and up to 12 weeks
  Functional Oral Intake Scale (FOIS) with a score range of 1( no oral intake) to 7 (Total oral diet with no restrictions).
Nutritional status | Baseline and up to 12 weeks
  The modified Mini Nutritional Assessment Scale-Short Form (MNA-SF). The total score range from 0 to 14, where a score <8 indicates malnutrition, 8-11 indicates risk of malnutrition, and >11 indicates no malnutrition.
Tongue strength and endurance | Baseline and up to 12 weeks
  Iowa Oral Performance Instrument (IOPI).
Intervention progress _ swallow difficulty | During two therapy sessions per week in 12 weeks.
  Self-reported swallowing difficulty of saliva, liquid and food (100 mm VAS scale (left side = no difficulties and right side = unable to swallow).
Intervention progress_ intensity | During two therapy sessions per week in 12 weeks.
  Self-perceived effort from 0 (at rest) to 10 (extremely hard).
Intervention progress _ Swallow ability | During two therapy sessions per week in 12 weeks.
  Records on observed number of successful/unsuccessful swallows.

OTHER OUTCOMES:
Demand for the intervention by the target group | Though study completion, an average of three years.
  Records of recruitment/attrition rates.
Intervention functionality | Though study completion, an average of three years.
  Records of numbers of complete/incomplete therapy sessions.
Intervention adaptations | During two therapy sessions per week in 12 weeks.
  Records on any adaptations (minor or major modifications, addition of new components, or deletions of a component) in the intervention model of the ACT-ING program during therapy. For any adaptations, 'what', 'how' and 'why' are recorded.
Determinants for delivering the ACT-ING program by practitioners | Up to 12 weeks.
  Semi-structured interview based on the Theoretical Domains Framework

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided